CLINICAL TRIAL: NCT04664322
Title: High-flow Oxygen Therapy Versus Non-invasive Ventilation: a Randomised Physiological Cross-over Study of Alveolar Recruitment in Acute Respiratory Failure
Brief Title: High-flow Oxygen Therapy vs Non-invasive Ventilation: Comparison of Alveolar Recruitment in Acute Respiratory Failure
Acronym: IRAvista
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A00122-47; CPP-CS 001/2015 (Other: CPP Nord Ouest 1)
Record Dates: First submitted 2020-11-19; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Acute Respiratory Failure With Hypoxia
Keywords: alveolar recruitment; electrical impedance tomography; non-invasive ventilation; high-flow nasal cannula oxygen therapy; hypoxemic acute respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NIV/HFNC: patients receiving non-invasive ventilation than high flow nasal canulae oxygen therapy
  Interventions: Device: non invasive ventilation and high flow nasal canulae oxygen therapy
- HFNC/NIV: patients receiving high flow nasal canulae oxygen therapy than non-invasive ventilation
  Interventions: Device: non invasive ventilation and high flow nasal canulae oxygen therapy

INTERVENTIONS:
Device: non invasive ventilation and high flow nasal canulae oxygen therapy — patients with hypoxemic acute respiratory failure received alternatively non invasive ventilation and high flow nasal canulae oxygen therapy

SUMMARY:
This physiological study showed an increase in regional ventilation with NIV but no difference in alveolar recruitment as compared to HFNC in patients with hypoxemic ARF. Although NIV provided better oxygenation than HFNC, the effect on lung volumes could explain the potentially deleterious effect of NIV in hypoxemic ARF, reinforcing the recently developed concept of patient self-inflicted lung injury.

DETAILED DESCRIPTION:
Background: High-flow nasal cannula (HFNC) oxygen therapy has recently shown clinical benefits in hypoxemic acute respiratory failure (ARF) patients, while the interest of non-invasive ventilation (NIV) remains debated. The primary endpoint was to compare alveolar recruitment using global end-expiratory electrical lung impedance (EELI) between HFNC and NIV. Secondary endpoints compared regional EELI, lung volumes (global and regional tidal volume variation (TV)), respiratory parameters, hemodynamic tolerance, dyspnea and patient comfort between HFNC and NIV, relative to face mask (FM).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred in ICU
* with hypoxemic acute respiratory failure due to a community acquired pneumonia confirmed by chest X ray,
* with PaO2 < 60mmHg in ambient air, without hypercapnia (PaCO2 < 45 mmHg),
* requiring more than 6L/min of O2 on admission with high concentration FM, and justifying HFNC or NIV for the attending ICU physician

Exclusion Criteria:

* cardiogenic pulmonary oedema,
* moderate to severe underlying respiratory disease including COPD (chronic obstructive pulmonary disease)
* contraindication to or failure of previous NIV or HFNC with the need for immediate invasive ventilation
* pregnant or breast-feeding women
* carrier of an implantable defibrillator or pacemaker
* body mass index (BMI)>50 kg/m2
* with cutaneous lesion next to the positioning zone of the Pulmovista® (Dräger, Lübeck, Germany) belt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults referred in ICU
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
global EELI | after 5 minutes of stable breathing with the oxygenation technic
  measurement of global end respiratory lung impedance with non invasive ventilation vs with high flow nasal canulae oxygen therapy, standard unit

SECONDARY OUTCOMES:
ROI EELI | after 5 minutes of stable breathing with the oxygenation technic
  measurement of regional of interest (ROI) end respiratory lung impedance with non invasive ventilation vs with high flow nasal canulae oxygen therapy, standard unit
global TV | after 5 minutes of stable breathing with the oxygenation technic
  measurement of global tidal variation (TV) with non invasive ventilation vs with high flow nasal canulae oxygen therapy, standard unit
ROI TV | after 5 minutes of stable breathing with the oxygenation technic
  measurement of regional tidal variation with non invasive ventilation vs with high flow nasal canulae oxygen therapy, standard unit

CONTACTS AND LOCATIONS:
Overall Officials: Christophe GIRAULT, MD, Study Director — Medical Intensive Care Department, Rouen University Hospital, F-76000 Rouen, France

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP
Time Frame: from the first patient enrollment ( 02/22/2016) to publication
Access Criteria: Excel database was shared with biostatisticians for statistical analysis